CLINICAL TRIAL: NCT00004689
Title: Phase II Study of Amithiozone (Thiacetazone) for Patients With Mycobacterium Avium Complex Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Jewish Health (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 199/13311; NJCIRM-HS-750; NJCIRM-FDR000812
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-02

CONDITIONS: Mycobacterium Avium-intracellulare Infection
Keywords: bacterial infection; immunologic disorders and infectious disorders; mycobacterium avium infection; mycobacterium infection; rare disease
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; Bacterial Infections; Immune System Diseases; Communicable Diseases; Mycobacterium Infections; Rare Diseases | interventions — Thioacetazone; Clarithromycin; Ethambutol; Rifampin; Streptomycin

INTERVENTIONS:
Drug: amithiozone
Drug: clarithromycin
Drug: ethambutol
Drug: rifampin
Drug: streptomycin

SUMMARY:
OBJECTIVES: I. Determine the bacteriological activity of amithiozone against Mycobacterium avium complex (MAC) pulmonary disease.

II. Define the ability of amithiozone to improve clinical outcomes in patients with MAC infection.

III. Determine the safety and tolerance of amithiozone with chronic dosing in these patients.

IV. Assess the contribution of clarithromycin, streptomycin, rifampin, ethambutol, kanamycin, and amithiozone in the treatment of pulmonary MAC infection.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: The is a randomized, open label study. All patients receive a core regimen of clarithromycin and streptomycin. Patients are randomized into two treatment arms. Arm I patients receive rifampin and ethambutol. Arm II patients receive amithiozone.

Patients are followed for one year to detect any relapse or other complications.

Patients not eligible for this randomized study may be entered on a short open label study with amithiozone.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Progressive pulmonary disease due to Mycobacterium avium complex (MAC) as defined by: Three of more sputum culture(s) positive for MAC Change in serial chest roentgenograms consistent with active mycobacterial disease over a 12 week period No other obvious cause of pulmonary disease
* Patients must have organisms that are: Susceptible to amithiozone AND Susceptible or moderately susceptible to the combination of rifampin and ethambutol, and to clarithromycin and streptomycin

--Prior/Concurrent Therapy--

* No likelihood of resectional thoracic surgery within 24 weeks of evaluation

--Patient Characteristics--

* Age: 18 and over
* Performance status: Not specified
* Hematopoietic: Not specified
* Hepatic: Bilirubin less than 3 times normal SGOT/SGPT less than 3 times normal Alkaline phosphatase less than 3 times normal
* Renal: Creatinine clearance at least 30 mL/min
* Cardiovascular: No New York Heart Association class III or IV heart failure
* Other: No optic disease that precludes the use of ethambutol No hypersensitivity to rifampin, ethambutol, clarithromycin, streptomycin, or amithiozone HIV negative Not pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 1991-01; Study Completion 1998-09

CONTACTS AND LOCATIONS:
Overall Officials: Charles Arthur Peloquin, Study Chair — National Jewish Health